CLINICAL TRIAL: NCT01120353
Title: Childhood Cancer Survivor Study
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other); Nationwide Children's Hospital (Other); M.D. Anderson Cancer Center (Other); University of Southern California (Other); Children's Hospital Medical Center, Cincinnati (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CCSS; U24CA055727 (NIH); R03CA169150 (NIH); R01CA134722 (NIH); R01CA136783 (NIH); R01CA132899 (NIH); R01CA187397 (NIH); R01CA175231 (NIH); R21CA202210 (NIH); R21CA198641 (NIH); NCI-2021-05717 (Registry Identifier: NCI)
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Childhood cancer; Young Children; Adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, saliva and second tumor specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer survivors: Survivors of cancer, diagnosed under 21 years of age, between 1970 and 1999 This project will study children and young adults exposed to specific therapeutic modalities, including radiation, chemotherapy, and/or surgery, for an increased risk of late-occurring events associated with excess mortality and morbidity.
- Sibling Controls: A group of sibling controls will be identified to provide: (1) the ability to make direct comparisons with the survivors, (2) data on outcomes in a non-cancer population, and (3) additional comparison group to determine consistency of findings between data sources.

SUMMARY:
The Childhood Cancer Survivor Study (CCSS) will investigate the long-term effects of cancer and its associated therapies. A retrospective cohort study will be conducted through a multi-institutional collaboration, which will involve the identification and active follow-up of a cohort of approximately 50,000 survivors of cancer, diagnosed before 21 years of age, between 1970 and 1999 and 10,000 sibling controls. This project will study children and young adults exposed to specific therapeutic modalities, including radiation, chemotherapy, and/or surgery, who are at increased risk of late-occurring adverse health outcomes. A group of sibling controls will be identified and data collected for comparison purposes.

DETAILED DESCRIPTION:
The study will focus on the following objectives:

* Characterize survivors' health with respect to disease- and treatment-related factors.
* Investigate the consequences of various intensities of exposure to chemotherapy and/or radiation on health outcomes (e.g., cardiovascular, reproductive, second cancers, etc…).
* Compare the mortality experience of survivors with the general population.
* Characterize the health-related behaviors, patterns of medical care, and medical follow-up needs of survivors.
* Describe patterns of familial aggregation of cancer, including known (and variations of) cancer family syndromes.
* Collect and store biologic samples (saliva, blood, second tumor tissue) to correlate with health outcomes and use for future research.

ELIGIBILITY:
Inclusion Criteria:

Initial Cohort:

* Five-year survival following diagnosis of leukemia, lymphoma, CNS tumor, bone tumor, Wilms tumor, neuroblastoma, or soft tissue sarcoma before age 21 years between January 1, 1970 and December 31, 1986 at one of participating centers.

Expanded cohort:

* Five-year survival following diagnosis of leukemia, lymphoma, CNS tumor, bone tumor, kidney tumor, neuroblastoma, or rhabdomyosarcoma before age 21 years between January 1, 1987 and December 31, 1999 at one of participating centers.
* English- or Spanish-speaking and living in the U.S. or Canada at the time of diagnosis.

Exclusion Criteria:

* Diagnosis of non-malignant tumors (i.e., Langerhans cell histiocytosis, meningioma, craniopharyngioma, etc.) treated with radiation and/or chemotherapy.
* Non-English speaking or residence outside the US or Canada.

Sibling Controls:

* For comparison purposes, a group of sibling controls will be identified to represent a stratified random sample based on the distribution of survivors with regard to cancer diagnosis, age, sex, race, and geographic location.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed with cancer between January 1, 1970 and December 31, 1999 at one of the participating centers noted below or identified as sibling control.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 1995-01-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
To characterize survivors' health outcomes with respect to disease-, treatment, and genetic-related factors. | 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregory T. Armstrong, MD, MSCE, Principal Investigator — St. Jude Children's Research Hospital
Locations (31):
- United States (30):
  - University of Alabama at Birmingham/Children's of Alabama, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California-Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California-San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University/Children's Health Care of Atlanta, Atlanta, Georgia
  - Ana & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University/Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan/Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals & Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis Children's Hospital/The Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial-Sloan Kettering Cancer Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Alberts NM, Leisenring W, Whitton J, Stratton K, Jibb L, Flynn J, Pizzo A, Brinkman TM, Birnie K, Gibson TM, McDonald A, Ford J, Olgin JE, Nathan PC, Stinson JN, Armstrong GT. Characterization of chronic pain, pain interference, and daily pain experiences in adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Pain. 2024 Nov 1;165(11):2530-2543. doi: 10.1097/j.pain.0000000000003284. Epub 2024 Jul 9. PMID 38981063
- [Derived] Wilson CL, Bjornard KL, Partin RE, Kadan-Lottick NS, Nathan PC, Oeffinger KC, Hayashi RJ, Hyun G, Armstrong GT, Leisenring WM, Howell RM, Yasui Y, Dixon SB, Ehrhardt MJ, Robison LL, Ness KK. Trends in physical functioning in acute lymphoblastic leukemia and non-Hodgkin lymphoma survivors across three decades. J Cancer Surviv. 2025 Apr;19(2):496-506. doi: 10.1007/s11764-023-01483-1. Epub 2023 Nov 8. PMID 37938431
- [Derived] Chen C, Qin N, Wang M, Dong Q, Tithi SS, Hui Y, Chen W, Wu G, Kennetz D, Edmonson MN, Rusch MC, Thrasher A, Easton J, Mulder HL, Song N, Plonski NM, Shelton K, Im C, Ehrhardt MJ, Nichols KE, Leisenring WM, Stratton KL, Howell R, Yasui Y, Bhatia S, Armstrong GT, Ness KK, Hudson MM, Zhang J, Wang H, Srivastava DK, Robison LL, Wang Z. Cancer germline predisposing variants and late mortality from subsequent malignant neoplasms among long-term childhood cancer survivors: a report from the St Jude Lifetime Cohort and the Childhood Cancer Survivor Study. Lancet Oncol. 2023 Oct;24(10):1147-1156. doi: 10.1016/S1470-2045(23)00403-5. PMID 37797633
- [Derived] Mulrooney DA, Hyun G, Ness KK, Ehrhardt MJ, Yasui Y, Duprez D, Howell RM, Leisenring WM, Constine LS, Tonorezos E, Gibson TM, Robison LL, Oeffinger KC, Hudson MM, Armstrong GT. Major cardiac events for adult survivors of childhood cancer diagnosed between 1970 and 1999: report from the Childhood Cancer Survivor Study cohort. BMJ. 2020 Jan 15;368:l6794. doi: 10.1136/bmj.l6794. PMID 31941657
- [Derived] Ness KK, Hudson MM, Jones KE, Leisenring W, Yasui Y, Chen Y, Stovall M, Gibson TM, Green DM, Neglia JP, Henderson TO, Casillas J, Ford JS, Effinger KE, Krull KR, Armstrong GT, Robison LL, Oeffinger KC, Nathan PC. Effect of Temporal Changes in Therapeutic Exposure on Self-reported Health Status in Childhood Cancer Survivors. Ann Intern Med. 2017 Jan 17;166(2):89-98. doi: 10.7326/M16-0742. Epub 2016 Nov 8. PMID 27820947
- [Derived] Patterson BC, Chen Y, Sklar CA, Neglia J, Yasui Y, Mertens A, Armstrong GT, Meadows A, Stovall M, Robison LL, Meacham LR. Growth hormone exposure as a risk factor for the development of subsequent neoplasms of the central nervous system: a report from the childhood cancer survivor study. J Clin Endocrinol Metab. 2014 Jun;99(6):2030-7. doi: 10.1210/jc.2013-4159. Epub 2014 Feb 25. PMID 24606096
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Long-Term Follow-Up Study — http://ltfu.stjude.org/
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols